CLINICAL TRIAL: NCT01529450
Title: A Pilot Open-Label Study to Examine the Safety and Efficacy of Oral LDE225 in Patients With Locally Advanced or Metastatic Basal Cell Carcinoma Who Have Been Previously Treated With Non-LDE225 Smoothened Inhibitor(s)
Brief Title: Pilot LDE225 in Locally Advanced or Metastatic BCC + Previously Tx Non-LDE225 Smoothened Inhibitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Chang (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Anne Chang, Assistant Professor of Dermatology, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKIN0009; SU-09022011-8371 (Other: Stanford University); 21759 (Other: Stanford IRB)
Record Dates: First submitted 2011-10-11; First posted 2012-02-08 (Estimated); Results first posted 2016-11-02 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Basal Cell Carcinoma
Keywords: basal cell carcinoma, sonidegib, smoothened inhibitor, hedgehog
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Refractory Group (Active Comparator): Patients previously treated with non-LDE225 Smo inhibitor who were refractory.
  Interventions: Drug: LDE225
- Resistance Developed Group (Active Comparator): Patients previously treated with non-LDE225 Smo inhibitor who were initially responsive but became resistant with progressive disease.
  Interventions: Drug: LDE225

INTERVENTIONS:
Drug: LDE225 — 800-mg (4 200-mg capsules/day) capsule
  Other Names: NVP-LDE225

SUMMARY:
This is a prospective single-center, open label, pilot study to investigate the safety and efficacy of LDE225 in patients with locally advanced or metastatic basal cell carcinoma.

Primary Objectives:

• To explore the effects of oral LDE225 on the Progression Free Survival (PFS) of individuals with locally advanced or metastatic BCC who have been previously treated with a non-LDE225 Smo inhibitor.

Secondary Objectives:

* To evaluate the effect of oral LDE225 on tumor tissue biomarkers of BCC activation (Gii 1, 2, Patched 1,2 and Ki67) in individuals which are non-na"ive to Smo inhibitors other than LDE225, at baseline and at end-of-treatment
* To describe adverse effects of oral LDE225 in individuals with a history of non-LDE225 Smo inhibitor usage
* To assess the overall survival rates of individuals with locally advanced BCC or metastatic BCC who have previously taken a non-LDE225 Smo inhibitor after treatment with LDE225

DETAILED DESCRIPTION:
This is a prospective single-center, open label, pilot study to investigate the safety and efficacy of LDE225 in patients with locally advanced or metastatic basal cell carcinoma.

Primary Objectives:

• To explore the effects of oral LDE225 on the Progression Free Survival (PFS) of individuals with locally advanced or metastatic BCC who have been previously treated with a non-LDE225 Smo inhibitor.

Secondary Objectives:

* To evaluate the effect of oral LDE225 on tumor tissue biomarkers of BCC activation (e.g. Gli and Ki67) in individuals which are non-naive to Smo inhibitors other than LDE225, at baseline and at end-of-treatment
* To describe adverse effects of oral LDE225 in individuals with a history of non-LDE225 Smo inhibitor usage

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Histologically documented diagnosis of basal cell carcinoma deemed to be locally advanced or metastatic who have previously received a non-LDE225 Smo inhibitor.
3. World Health Organization (WHO) performance status <= 2
4. At least one measurable site of disease (as defined by Response Evaluation Criteria in Solid Tumors), or other disease specific response assessment criteria, as appropriate. State age restriction and/or gender/race-ethnic restrictions.
5. Patients with adequate bone marrow, liver and renal function, as specified below:

   * Absolute Neutrophil Count (ANC) >= 1.5 x 10^9/L
   * Hemoglobin (Hgb) >= 9 g/dL
   * Platelets >= 80 x 10^9/L
   * Serum total bilirubin <= 1.5 x upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 2.5 x ULN or <= 5 x ULN if liver metastases are present
   * Plasma creatine phosphokinase (CK) < 1.5 x ULN
   * Serum creatinine <= 1.5 x ULN or 24-hour clearance >= 50ml/min
6. Written informed consent obtained prior to any screening procedures

Exclusion Criteria:

1. Patients who have had major surgery within 4 weeks of initiation of study medication.
2. Patients with concurrent uncontrolled medical conditions that may interfere with their participation in the study or potentially affect the interpretation of the study data.

   State restrictions regarding use of other Investigational Agents.
3. Patients unable to take oral drugs or with lack of physical integrity of the upper gastrointestinal tract or known malabsorption syndromes.

   State exclusion requirements due to co-morbid disease or incurrent illness, as needed.
4. Patients who have previously been treated with systemic LDE225.
5. Patients who have neuromuscular disorders (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy) or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis, such as 3-hydroxy-3-methylglutaryl-coenzyme A (HMG CoA) inhibitors (statins), clofibrate and gemfibrozil, and that cannot be discontinued at least 2 weeks prior to starting LDE225 treatment. If it is essential that the patient stays on a statin to control hyperlipidemia, only pravastatin may be used with extra caution.

   b) Patients who are planning on embarking on a new strenuous exercise regimen after initiation of study treatment. Note: Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided whilst on LDE225 treatment.
6. Patients who have taken part in an experimental drug study within 4 weeks of initiating treatment with LDE225.
7. Patients who are receiving other anti-neoplastic therapy (e.g. chemotherapy, targeted therapy or radiotherapy) concurrently or within 2 weeks of starting treatment with LDE225.
8. Patients who are receiving treatment with medications known to be moderate and strong inhibitors or inducers of cytochrome (CYP)3A4/5 or drugs metabolized by CYP2B6 or CYP2C9 that have narrow therapeutic index, and that cannot be discontinued before starting treatment with LDE225. Medications that are strong CYP3A4/5 inhibitors should be discontinued at least 7 days and strong CYP3A/5 inducers for at least 2 weeks prior to starting treatment with LDE225.
9. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 5 mIU/mL).

10 Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method. Adequate barrier methods of contraception include:

* Diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent.
* Reliable contraception should be maintained throughout the study and for 3 months after study drug discontinuation.

  11 Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Chang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Danial C, Sarin KY, Oro AE, Chang AL. An Investigator-Initiated Open-Label Trial of Sonidegib in Advanced Basal Cell Carcinoma Patients Resistant to Vismodegib. Clin Cancer Res. 2016 Mar 15;22(6):1325-9. doi: 10.1158/1078-0432.CCR-15-1588. Epub 2015 Nov 6. PMID 26546616

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Refractory Group | Resistance Developed Group
Started | 3 | 8
Completed | 3 | 6
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: Participants with evaluable data are included for Baseline Characteristics
Groups:
- Total: Total of all reporting groups
Arm/Group | Refractory Group | Resistance Developed Group | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (24) | 54 (9) | 57 (15)
Gender [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 9
Size of disease by RECIST criteria [Mean (Standard Deviation); unit: centimeters] | 3.8 (1.3) | 4.2 (2.4) | 4.0 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) of All Participants
Time Frame: End of treatment or at time of disease progression (up to 58 weeks)
Population: Progression is defined using RECIST version 1.0 as a 20% increase in the sum of the longest diameter of target lesions, or a measureable increase in a non-target lesion or the appearance of new lesion.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Refractory Group | Resistance Developed Group
Number analyzed (Participants) | 3 | 6
weeks | 6 [3 to 12] | 36 [14 to 58]

2. Secondary Outcome: Molecular Markers Associated With Clinical Response
Description: Following consent, historical biopsy samples were analyzed for molecular markers associated with clinical response. Tumors were analyzed and present of Smooth mutation (SMO [genetic changes which influence Ki 67 and Gli levels]). was determined. The number of participants with and without SMO were reported by clinical outcome (SD = stable disease; PD = progressive disease).
Time Frame: Assessed on day 1
Population: Participants with tissue available for screening were analyzed.
Measure: Number; unit: participants
Groups:
- All Participants: Participants received LDE225: 800-mg (4 200-mg capsules/day) capsule
Arm/Group | All Participants
Number analyzed (Participants) | 7
participants
  SMO Present (outcome SD) | 1
  SMO absent (outcome SD) | 1
  SMO Present (outcome PD) | 4
  SMO absent (outcome PD) | 1

ADVERSE EVENTS:
Description: Participants with evaluable data are included for Adverse Events
Arm/Group | Refractory Group | Resistance Developed Group
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Refractory Group (N=3) | Resistance Developed Group (N=6)
Altered mental status (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Refractory Group (N=3) | Resistance Developed Group (N=6)
palpitations (Cardiac disorders) | 0 | 1 — Grade 1
ear canal stenosis (Ear and labyrinth disorders) | 1 | 0 — Grade 1
ear drainage (Ear and labyrinth disorders) | 1 | 0 — Grade 1
hearing loss (Ear and labyrinth disorders) | 1 | 0 — Grade 2
appetite decrease (Gastrointestinal disorders) | 1 | 0 — Grade 1
dehydration (Gastrointestinal disorders) | 0 | 1 — Grade 4
diarrhea (Gastrointestinal disorders) | 1 | 0 — Grade 1
nausea (Gastrointestinal disorders) | 0 | 2 — Grade 4
taste disturbance (Gastrointestinal disorders) | 0 | 1 — Grade 1
vomit (Gastrointestinal disorders) | 1 | 0 — Grade 1
weight loss (General disorders) | 1 | 0 — Grade 2
candidiasis (Infections and infestations) | 1 | 0 — Grade 2
ecchymosis (Injury, poisoning and procedural complications) | 0 | 1 — Grade 2
laceration (Injury, poisoning and procedural complications) | 0 | 1 — Grade 2
elevated creatine kinase (Investigations) | 0 | 1 — Grade 1
hip fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 — Grade 4
muscle cramps (Musculoskeletal and connective tissue disorders) | 0 | 4 — Grade 1
restless arms and legs (Musculoskeletal and connective tissue disorders) | 0 | 1 — Grade 1
rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 — Grade 4
neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Grade 2
altered mental status (Nervous system disorders) | 0 | 1 — Grade 4
migraine (Nervous system disorders) | 1 | 0 — Grade 1
somnolence (Nervous system disorders) | 1 | 0 — Grade 1
agitation (Psychiatric disorders) | 0 | 1 — Grade 1
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No